CLINICAL TRIAL: NCT00715780
Title: Observational Safety and Efficacy Study in Subjects Using Insulin for the Treatment of Type 2 Diabetes Mellitus Failing on Oral Anti-diabetic Agents
Brief Title: Observational Study to Evaluate Safety and Efficacy of Insulin Therapy in Type 2 Diabetes Mellitus Subjects Failing on Oral Anti-diabetic Agents
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3615
Record Dates: First submitted 2008-07-14; First posted 2008-07-15 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin; biphasic human insulin 30; Insulin, Isophane; Insulin Aspart; insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: soluble human insulin; Drug: biphasic human insulin; Drug: insulin NPH; Drug: insulin aspart; Drug: biphasic insulin aspart; Drug: insulin detemir

INTERVENTIONS:
Drug: soluble human insulin — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Other Names: Actrapid®
Drug: biphasic human insulin — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
Drug: insulin NPH — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
Drug: insulin aspart — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
Drug: biphasic insulin aspart — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
Drug: insulin detemir — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate the incidence of major hypoglycaemic episodes and other adverse events, and to evaluate efficacy while using insulin under normal clinical practice conditions. The switch from OAD treatment to insulin therapy will be determined by physician.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 12 months and currently receiving oral anti-diabetic (OAD) treatment, whether single or combination, for at least 3 months before this study
* Insulin naive
* Poor glycaemic control on OADs and decided by the physician to start insulin therapy

Exclusion Criteria:

* Type 1 diabetes patients
* Patients who are unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for the final visit
* Patients with a hypersensitivity to insulin or to any of the excipients
* Patient groups not approved in the product label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic patients
Sampling Method: Probability Sample
Enrollment: 1667 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Incidence of major hypoglycaemic episodes | during 26 weeks of insulin therapy

SECONDARY OUTCOMES:
Frequency and type of hypoglycaemic episodes | during 26 weeks of insulin therapy
Frequency and type of adverse events | during 26 weeks of insulin therapy
Frequency and type of adverse drug reactions | during 26 weeks of insulin therapy
Change in HbA1c from baseline | during 26 weeks of insulin therapy
Change in PPG from baseline | during 26 weeks of insulin therapy
Change in FPG from baseline | during 26 weeks of insulin therapy
Subjects' insulin treatment satisfaction | during 26 weeks of insulin therapy
Physicians' satisfaction with insulin therapy | during 26 weeks of insulin therapy
Weight change | at the end of the study
Percentage of patients reaching the target of HbA1c less than 7.5% | at the end of the study
Percentage of patients reaching the target of HbA1c less than 7% | at the end of the study
Percentage of patients reaching the target of HbA1c less than 6.5% | at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Jakarta, Indonesia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com